CLINICAL TRIAL: NCT05618808
Title: A Phase 2, Multicenter, Randomized, Open-Label, Active-Control Study of REGN9933, a Factor XI Monoclonal Antibody, for Prevention of Venous Thromboembolism After Elective, Unilateral, Total Knee Arthroplasty
Brief Title: A Trial to Learn How Well REGN9933 Works for Preventing Blood Clots After Knee Replacement Surgery in Adult Participants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R9933-DVT-2230; 2022-501470-18-00 (Other: EU CT)
Record Dates: First submitted 2022-11-08; First posted 2022-11-16 (Actual); Results first posted 2025-07-16 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Venous Thromboembolism
Keywords: Anti-factor XI (FXI) monoclonal antibody; Deep Vein Thrombosis; Unilateral total knee arthroplasty (TKA),
MeSH Terms: conditions — Venous Thromboembolism; Venous Thrombosis | interventions — Enoxaparin; apixaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- REGN9933 (Experimental): REGN9933 will be administered by intravenous (IV) infusion
  Interventions: Drug: REGN9933
- Enoxaparin (Active Comparator): Enoxaparin will be administered by subcutaneous (SC) administration
  Interventions: Drug: Enoxaparin
- Apixaban (Active Comparator): Apixaban will be administered orally twice a day
  Interventions: Drug: Apixiban

INTERVENTIONS:
Drug: REGN9933 — Participants will receive a single dose of REGN9933 by IV infusion
  Arms: REGN9933
Drug: Enoxaparin — Participants will receive enoxaparin by SC administration daily through the time of venography (or day 12, whichever is earlier)
  Other Names: Lovenox
  Arms: Enoxaparin
Drug: Apixiban — Participants will receive apixaban orally twice a day through the time of venography (or day 12, whichever is earlier)
  Other Names: Eliquis
  Arms: Apixaban

SUMMARY:
The primary objective of the study is to evaluate the efficacy of REGN9933 for the prevention of venous thromboembolism (VTE) after unilateral total knee arthroplasty (TKA), compared to enoxaparin

The secondary objectives of the study are:

* To evaluate the bleeding risk (ie, major and clinically relevant non-major [CRNM] bleeding) of REGN9933 after unilateral TKA through time of venography, compared to enoxaparin
* To assess overall safety and tolerability of REGN9933 in participants undergoing TKA
* To evaluate the efficacy of REGN9933 in prevention of clinically relevant VTE, compared to enoxaparin
* To evaluate the efficacy of REGN9933 in prevention of deep venous thrombosis (DVT) detected by venography, compared to enoxaparin
* To evaluate the pharmacokinetics (PK) of REGN9933 after single intravenous (IV) administration
* To assess pharmacodynamic (PD) effects of REGN9933 on intrinsic and extrinsic coagulation pathways
* To assess immunogenicity following a single dose of REGN9933 over time
* To compare the efficacy of enoxaparin and apixaban in prevention of VTE after unilateral TKA

ELIGIBILITY:
Key Inclusion Criteria:

1. Undergoing elective unilateral TKA
2. Has a body weight ≤130 kg at screening visit
3. Is judged by the investigator to be in good health based on medical history, physical examination, vital sign measurements, and Electrocardiograms (ECG) performed at screening and/or prior to administration of initial dose of study drug
4. Is in good health based on laboratory safety testing obtained during the screening period as described in the protocol

Key Exclusion Criteria:

1. History of bleeding in the past 6 months requiring hospitalization or transfusion; history of intracranial or intraocular bleeding, excessive operative or post-operative bleeding, and traumatic spinal or epidural anesthesia; history of bleeding diathesis.
2. History of thromboembolic disease or thrombophilia
3. History of major surgery, including brain, spinal, or ocular, within approximately the past 6 months.
4. History of major trauma within approximately the past 6 months.
5. Hospitalized (>24 hours) for any reason within 30 days of the screening visit
6. Using the Modification of Diet in Renal Disease equation, has an estimated glomerular filtration rate as described in the protocol

Note: Other protocol-defined Inclusion/ Exclusion Criteria apply

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 373 (Actual)
Dates: Start 2023-05-24 (Actual); Primary Completion 2024-05-27 (Actual); Study Completion 2024-05-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (16):
- Ziekenhuis Oost-Limburg- Campus Sint-Jan, Genk, Limburg, Belgium
- MBAL Heart and Brain Hospital, Pleven, Bulgaria
- Durham Bone and Joint Specialists, Ajax, Ontario, Canada
- Hungary (2):
  - MAV Korhaz es Rendelointezet Szolnok, Szolnok, Jász-Nagykun-Szolnok
  - Department of Orthopedics, Somogy County Mór Kaposi Teaching Hospital, Kaposvár
- Latvia (4):
  - Liepaja Regional Hospital, Liepāja
  - Vidzemes Hospital, Riga
  - Riga's 2nd Hospital, Riga
  - Hospital of Traumatology and Orthopaedics, Riga
- Lithuania (3):
  - Lietuvos Sveikatos Mokslu Universiteto Ligonine Kauno Klinik, Kaunas, Kaunas County
  - Klaipeda University Hospital, Klaipėda, Klaipėda County
  - Lietuvos Sveikatos Mokslu Universiteto Kauno Ligoninė, Kaunas
- Poland (4):
  - Specjalistyczny Szpital im. E. Szczeklika w Tarnowie, Tarnów, Lesser Poland Voivodeship
  - SP ZOZ Centralny Szpital Kliniczny UM w Lodzi, Lodz
  - Samodzielny Publiczny Szpital Kliniczny nr 4 w Lublinie, Lublin
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej w Radzyniu Podlaskim, Radzyń Podlaski

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication, has made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry), has the legal authority to share the data, and has ensured the ability to protect participant privacy.
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/

REFERENCES:
- [Derived] Weitz JI, Kithcart AP, O'Brien MP, Levy O, Marin E, Onisko M, Mohammadi KA, Li D, Meagher KA, Chang HH, Olenchock BA, Gutstein DE, Segers A, Roberts RS, Bonaca MP, Raskob GE. Efficacy and safety of REGN9933A2 and REGN7508Cat for preventing postoperative venous thromboembolism (ROXI-VTE-I and ROXI-VTE-II): two randomised, open-label, phase 2 trials. Lancet. 2025 Nov 29;406(10519):2551-2563. doi: 10.1016/S0140-6736(25)02097-5. Epub 2025 Nov 8. PMID 41218619
- See also: Related Info — https://roxi-vte.com
- See also: A Plain Language Summary is available on TrialSummaries.com — https://www.trialsummaries.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 450 participants were screened for study eligibility, and 77 participants discontinued during the screening period. 373 participants met eligibility criteria and were randomized into 1 of 3 treatment groups.
Groups:
- REGN9933: REGN9933 was administered by intravenous (IV) infusion
- Enoxaparin: Enoxaparin was administered by subcutaneous (SC) administration
- Apixaban: Apixaban was administered orally twice a day
Period: Overall Study
Arm/Group | REGN9933 | Enoxaparin | Apixaban
Started (All randomized participants) | 123 | 125 | 125
Completed (Randomized participants who completed the study) | 120 | 124 | 122
Not Completed | 3 | 1 | 3
Not completed — Withdrawal by Subject | 3 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | REGN9933 | Enoxaparin | Apixaban | Total
Number analyzed (Participants) | 123 | 125 | 125 | 373
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.5 (7.73) | 66.6 (7.61) | 66.5 (7.69) | 66.5 (7.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 104 | 89 | 288
  Male | 28 | 21 | 36 | 85
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 4 | 9
  Not Hispanic or Latino | 120 | 121 | 121 | 362
  Unknown or Not Reported | 0 | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 123 | 125 | 125 | 373
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Confirmed, Adjudicated Venous Thromboembolism (VTE) (REGN9933 vs Enoxaparin)
Description: Composite endpoint that includes: asymptomatic deep DVT (deep venous thrombosis) detected by unilateral venography of the operated leg; confirmed symptomatic DVT of either leg; confirmed fatal or nonfatal pulmonary embolism (PE) including unexplained death for which PE cannot be ruled out
Time Frame: Through Day 12
Population: Randomized participants in the REGN9933 and enoxaparin arms that had either an evaluable venogram, a confirmed episode of venous thromboembolism, or both.
Measure: Number; unit: percentage of participants
Arm/Group | REGN9933 | Enoxaparin
Number analyzed (Participants) | 116 | 117
percentage of participants | 17.2 | 22.2
Statistical Analysis 1: Comparison: REGN9933 vs Enoxaparin; Test type: Superiority; Posterior Odds Ratio = 0.78, 90% CI 2-sided [0.47 to 1.32] — REGN9933 vs Enoxaparin; Bayesian Logistic Regression; "Confidence Interval" refers to "Credible Interval"

2. Secondary Outcome: Number of Participants With Major Bleeding and Clinically Relevant Non-major (CRNM) Bleeding
Description: International Society on Thrombosis and Hemostasis (ISTH) criteria for Major Bleeding and CRNM Bleeding as described in the protocol
Time Frame: Through Day 12
Population: Randomized participants that had either an evaluable venogram, a confirmed episode of venous thromboembolism, or both.
Measure: Count of Participants; unit: Participants
Arm/Group | REGN9933 | Enoxaparin | Apixaban
Number analyzed (Participants) | 116 | 117 | 113
Participants | 0 | 0 | 0

3. Secondary Outcome: Percentage of Participants With at Least One Treatment Emergent Adverse Event (TEAE)
Description: A TEAE is any untoward medical occurrence in a participant administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment.
Time Frame: Up to Day 75
Measure: Number; unit: percentage of participants
Arm/Group | REGN9933 | Enoxaparin | Apixaban
Number analyzed (Participants) | 123 | 125 | 125
percentage of participants | 22.0 | 20.8 | 24.8

4. Secondary Outcome: Percentage of Participants With Major VTE (REGN9933 vs Enoxaparin)
Description: Major VTE is a composite endpoint that includes: proximal DVT; confirmed symptomatic DVT of either leg; confirmed fatal or nonfatal PE including unexplained death for which PE cannot be ruled out
Time Frame: Through Day 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | REGN9933 | Enoxaparin
Number analyzed (Participants) | 116 | 117
percentage of participants | 0 | 2.6
Statistical Analysis 1: Comparison: REGN9933 vs Enoxaparin; Test type: Superiority; Posterior Odds Ratio = 0.44, 90% CI 2-sided [0.16 to 1.61] — REGN9933 vs Enoxaparin; Bayesian Logistic Regression; "Confidence Interval" refers to "Credible Interval"

5. Secondary Outcome: Percentage of Participants With DVT (REGN9933 vs Enoxaparin)
Description: DVT measured by venography of the operated leg
Time Frame: Through Day 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | REGN9933 | Enoxaparin
Number analyzed (Participants) | 116 | 117
percentage of participants | 17.2 | 22.2
Statistical Analysis 1: Comparison: REGN9933 vs Enoxaparin; Test type: Superiority; Posterior Odds Ratio = 0.79, 90% CI 2-sided [0.47 to 1.32] — REGN9933 vs Enoxaparin; Bayesian Logistic Regression; "Confidence Interval" refers to "Credible Interval"

6. Secondary Outcome: Total REGN9933 Concentrations in Serum
Description: The concentrations of REGN9933 over time were summarized by descriptive statistics by study arm for the overall population
Time Frame: Days 0.0625 (post-dose), 4, 9, 29, and 74
Population: All participants in the REGN9933 treatment group who received study drug and who had at least 1 non-missing result following the first dose of study drug and who were evaluable at time points specified for this outcome measure.
Measure: Mean (Standard Deviation); unit: milligrams/Liter (mg/L)
Arm/Group | REGN9933
Number analyzed (Participants) | 123
milligrams/Liter (mg/L)
  Day 0.0625 (post-dose) | 65.6 (18.2)
  Day 4: number analyzed (Participants) | 121
  Day 4 | 34.9 (9.65)
  Day 9: number analyzed (Participants) | 122
  Day 9 | 23.7 (7.15)
  Day 29: number analyzed (Participants) | 117
  Day 29 | 5.51 (3.47)
  Day 74: number analyzed (Participants) | 120
  Day 74 | 0.140 (0.107)

7. Secondary Outcome: Fold Change From Baseline in Activated Partial Thromboplastin Time (aPTT)
Description: aPTT was used to measure the anticipated anticoagulant effect of REGN9933. Fold change is based on the follow-up value/baseline value within an arm.
Time Frame: Days 1, 5, 10, 30, and 75
Population: All randomized participants who received any study drug and who had at least 1 non-missing pharmacodynamic (PD) result following the first dose of study drug and who were evaluable at time points specified for this outcome measure.
Measure: Mean (Standard Deviation); unit: Fold Change
Arm/Group | REGN9933 | Enoxaparin | Apixaban
Number analyzed (Participants) | 123 | 125 | 123
Fold Change
  Day 1: number analyzed (Participants) | 123 | 0 | 0
  Day 1 | 1.84 (0.245) |  |
  Day 5: number analyzed (Participants) | 121 | 125 | 123
  Day 5 | 2.26 (0.309) | 1.11 (0.143) | 1.16 (0.163)
  Day 10: number analyzed (Participants) | 122 | 124 | 121
  Day 10 | 2.17 (0.443) | 1.04 (0.114) | 1.10 (0.117)
  Day 30: number analyzed (Participants) | 119 | 115 | 119
  Day 30 | 1.56 (0.385) | 1.01 (0.149) | 1.04 (0.129)
  Day 75: number analyzed (Participants) | 120 | 123 | 122
  Day 75 | 1.01 (0.132) | 1.01 (0.119) | 1.03 (0.120)

8. Secondary Outcome: Fold Change From Baseline in Prothrombin Time (PT)
Description: PT is a measure of extrinsic and/or common pathway function. Fold change is based on the follow-up value/baseline value within an arm.
Time Frame: Days 1, 5, 10, 30, and 75
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Fold Change
Arm/Group | REGN9933 | Enoxaparin | Apixaban
Number analyzed (Participants) | 123 | 125 | 123
Fold Change
  Day 1: number analyzed (Participants) | 123 | 0 | 0
  Day 1 | 1.01 (0.075) |  |
  Day 5: number analyzed (Participants) | 121 | 125 | 123
  Day 5 | 0.96 (0.086) | 0.94 (0.064) | 1.02 (0.091)
  Day 10: number analyzed (Participants) | 122 | 124 | 121
  Day 10 | 0.95 (0.108) | 0.94 (0.073) | 1.00 (0.089)
  Day 30: number analyzed (Participants) | 119 | 115 | 119
  Day 30 | 0.99 (0.220) | 0.97 (0.122) | 0.99 (0.183)
  Day 75: number analyzed (Participants) | 120 | 123 | 122
  Day 75 | 0.94 (0.145) | 0.93 (0.092) | 0.94 (0.073)

9. Secondary Outcome: Number of Participants With Anti-REGN9933 Antibodies by Status
Description: Immunogenicity characterized by anti-drug antibody (ADA) status
Time Frame: Through Day 75
Population: All participants who received study drug REGN9933 and had at least 1 non-missing ADA result following the first dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | REGN9933
Number analyzed (Participants) | 119
Participants
  Negative | 118
  Pre-existing Immunoreactivity | 1
  Treatment-emergent (TE) Response | 0
  Treatment-boosted (TB) Response | 0

10. Secondary Outcome: Number of Participants With Treatment-Emergent or Treatment-Boosted Anti-REGN13335 Antibodies by Maximum Titer Level
Description: Immunogenicity characterized per drug molecule by ADA status
Time Frame: Through Day 75
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | REGN9933
Number analyzed (Participants) | 119
Participants
  Low (<1,000) | 0
  Moderate (1,000 to 10,000) | 0
  High (>10,000) | 0

11. Secondary Outcome: Percentage of Participants With Confirmed, Adjudicated VTE (Enoxaparin vs Apixaban)
Description: Asymptomatic deep DVT detected by unilateral venography of the operated leg; confirmed symptomatic DVT of either leg; confirmed fatal or nonfatal pulmonary embolism (PE) including unexplained death for which PE cannot be ruled out.
Time Frame: Through Day 12
Population: Randomized participants in the enoxaparin and apixaban arms that had either an evaluable venogram, a confirmed episode of venous thromboembolism, or both.
Measure: Number; unit: percentage of participants
Arm/Group | Enoxaparin | Apixaban
Number analyzed (Participants) | 117 | 113
percentage of participants | 22.2 | 12.4
Statistical Analysis 1: Comparison: Enoxaparin vs Apixaban; Test type: Superiority; Posterior Odds Ratio = 0.54, 90% CI 2-sided [0.32 to 0.95] — Enoxaparin vs Apixaban; Bayesian Logistic Regression; "Confidence Interval" refers to "Credible Interval"

ADVERSE EVENTS:
Time Frame: From date of signing informed consent form (ICF) up to end of study (approximately 105 days)
Arm/Group | REGN9933 | Enoxaparin | Apixaban
All-Cause Mortality (participants affected / at risk) | 0/123 | 0/125 | 0/125
Serious Adverse Events (participants affected / at risk) | 4/123 | 1/125 | 2/125
Other Adverse Events (participants affected / at risk) | 9/123 | 11/125 | 16/125
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | REGN9933 (N=123) | Enoxaparin (N=125) | Apixaban (N=125)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | REGN9933 (N=123) | Enoxaparin (N=125) | Apixaban (N=125)
Anaemia postoperative (Injury, poisoning and procedural complications) | 9 (9) | 11 (11) | 16 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2023-03-15): https://cdn.clinicaltrials.gov/large-docs/08/NCT05618808/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-07): https://cdn.clinicaltrials.gov/large-docs/08/NCT05618808/SAP_001.pdf